CLINICAL TRIAL: NCT02490540
Title: ANI and SPI Guided Intraoperative Analgesia in Patients Undergoing Neurosurgical Procedures Under General Anaesthesia
Brief Title: ANI and SPI Guided Intraoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Dr., University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201506S 38P
Record Dates: First submitted 2015-06-18; First posted 2015-07-07 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia
Keywords: opioids; analgesia; pain; anesthesia
MeSH Terms: conditions — Agnosia; Pain | interventions — Sufentanil; Anesthesiologists

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anesthesiologist quided analgesia (Experimental): Sufentanil anesthesiologist analgesia is based on anesthesiologist decision.
  Interventions: Drug: Sufentanil anesthesiologist analgesia
- ANI guided analgesia (Experimental): Sufentanil ANI analgesia based on ANI analgesia monitor figures.
  Interventions: Drug: Sufentanil ANI analgesia
- SPI guided analgesia (Experimental): Sufentanil SPI analgesia is based on the SPI analgesia monitor figures.
  Interventions: Drug: Sufentanil SPI analgesia

INTERVENTIONS:
Drug: Sufentanil SPI analgesia — Sufentanil is given based on SPI value in the SPI guided analgesia group. The targer SPI range is set indiviudally based on the initial value of SPI recorded 5 minutes after the induction of anesthesia plus 10 points. In the ANI group, Sufentanil is given based on the ANI value, the target ANI range is 50 - 70. Values lower than 49 for 1 minute indicate the need of administering further dose of opioid, sufentanil is given in the same dose as initially. In the anesthesiologist guided analgesia group, Sufentanil is administered in a standardized manner.
  Other Names: Sufentanil, SPI
  Arms: SPI guided analgesia
Drug: Sufentanil ANI analgesia — Sufentanil is given based on ANI analgesia monitor figures in the sufentanil ANI analgesia group. Targeted ANI range is 50 - 70. Figures lower than 49 for 1 minute indicate the need of administering further dose of opioid, sufentanil is given in the same dose as initially and flushed with 20 ml of saline. The next dose of opioid can be given in the earliest after 3 minutes interval, if indicated according to ANI monitoring. The doses are repeated up to achievement of the targeted range of analgesia (ANI). The last dose of opioid can be given no later than 15 minutes before the end of surgery.
  Other Names: Sufentanil, ANI
  Arms: ANI guided analgesia
Drug: Sufentanil anesthesiologist analgesia — Sufentanil is given based on the anesthesiologist decision in the sufentanil anesthesiologist analgesia group. Sufentanil is administered in 20 minute intervals in a standardized manner, the same dose as initially is given and flushed with 20 ml of saline. Indication for additional administration of opioid beyond this interval is 25 % increase of systemic arterial pressure over the baseline and/or 35% increase of heart rate over the baseline. The next dose of opioid can be given in the earliest after 3 minutes interval. The doses are repeated up to achievement of the haemodynamic stability. The last dose of opioid can be given no later than 15 minutes before the end of surgery.
  Other Names: Sufentanil, anesthesiologist
  Arms: Anesthesiologist quided analgesia

SUMMARY:
There is accumulating evidence that inappropriate analgesia is asssociated with increasing risk of perioperative complications. The aim of the study is to compare intraoperative analgesia guided according to different methods of intraoperative analgesia monitoring, ANI and SPI respectively.

DETAILED DESCRIPTION:
The Surgical Pleth Index (SPI) and ANI (Analgesia Nociception Index) has been developed for monitoring of adequacy of analgesia during surgery.

The investigators want to compare anesthesiologist guided intraoperative analgesia with intraoperative analgesia guieded by ANI or SPI.

The following hypotheses have been made:

1. Anesthesiologist guided analgesia will result in lower surgical stress
2. Anesthesiologist guided analgesia will result in more hemodynamic stability and faster recovery of the patient after anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled neurosurgical procedures under general anesthesia
* GCS 15
* ASA physical status I - III
* elective procedures with estimated duration 1 - 3 hours

Exclusion Criteria:

* Presence of non-sinus rhythm
* pacemaker
* planned postoperative ventilation
* procedures with planned awake intervals
* chronic pain with opioid medication
* opioid addiction
* epidural administration of local anaesthetic in combination with opioid
* corticosteroid use
* hormonal contraception
* chronic respiratory disease with known respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Cortisol serum level | End of surgery
  nmol/l

SECONDARY OUTCOMES:
Time to spontaneous ventilation | From the end of anesthesia up to two hours
  min
Time to extubation | From the end of anesthesia up to two hours
  min
Pain intensity at the time of departure from the operating theater | At the time of departure from the operating room, up to 30 min from the end of anesthesia
  Assessment of pain using verbal pain scale (range 0-4)
Pain intensity at recovery room admission | At the time of ICU/recovery room admission, up to 15 minutes after ICU/recovery admission
  Assessment of pain using verbal pain scale (range 0-4)
Mean pain intensity at the ICU/recovery room | From the admission to the ICU or recovery room up to 2 hours postoperatively
  Mean value of pain intensity score using verbal pain scale (range 0-4)
Postoperative respiratory complications | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Number of participants with postoperative respiratory complications
Sufentanil dose | From the beginning of anesthesia up to the end of anesthesia, an expacted average duration of 2 hours
  microgramms per hour
Pain intensity | 1st postoperative day
  Assessment of pain using verbal pain scale (range 0-4)
Pain intensity | 2nd postoperative day
  Assessment of pain using verbal pain scale (range 0-4)
Pain intensity | 3rd postoperative day
  Assessment of pain using verbal pain scale (range 0-4)
Number of doses of opioid analgesics | Until the end of the 3rd postoperative day
  The total number of doses of opioid analgesics during the 3 postoperative days
Number of doses of non-opioid analgesics | Until the end of the 3rd postoperative day
  The total number of doses of non-opioid analgesics during the 3 postoperative days
Time to achievement of normal end-tidal CO2 value | From the end of anesthesia up to two hours
  min
Length of postoperative hospital stay | From the day of surgery up to the end of hospital stay, an expected average of 2 weeks
  days

CONTACTS AND LOCATIONS:
Overall Officials: Vlasta Dostalova, MD, PhD, Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia